CLINICAL TRIAL: NCT06164535
Title: The Effects of Some Antihyperglycemic Drugs on Cognitive Function and Risk of Depression of Diabetic Patients
Brief Title: The Effects of DPPIs on Cognitive Function of Diabetic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Collaborators: Clinical Pharmacy Department, Faculty of Pharmacy, 6 October University (Unknown); Faculty of Medicine, Minia University (Unknown)
Responsible Party: Principal Investigator, Asmaa Abdelfattah Elsayed, Lecturer of clinical pharmacy, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BeniSuefU2023
Record Dates: First submitted 2023-11-30; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Cognitive Impairment
Keywords: Cognitive; DPP-4 inhibitors; Diabetes; Depression
MeSH Terms: conditions — Cognitive Dysfunction; Diabetes Mellitus; Depression | interventions — Control Groups; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: all patient information will be anonymized giving only corresponding numbers, which will be revealed by the PI after assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (Placebo Comparator): 35 patients will be given placebo (only adjust their drugs to control blood glucose level)
  Interventions: Drug: Control group
- DPPI Group (Experimental): 35 T2DM patients will be given DPP4Is once or twice daily
  Interventions: Drug: DPP-4 inhibitor group
- DPPI + metformin group (Experimental): 35 T2DM patients will be given DPP4Is + metformin once or twice daily
  Interventions: Drug: DPP-4 inhibitor + metformin group

INTERVENTIONS:
Drug: Control group — 35 T2DM patients will be given placebo (only adjust their drugs to control blood glucose level)
  Arms: Control Group
Drug: DPP-4 inhibitor group — 35 T2DM patients will be given DPP-4 I once or twice daily
  Arms: DPPI Group
Drug: DPP-4 inhibitor + metformin group — 35 T2DM patients will be given DPP-4 I + metformin once or twice daily
  Arms: DPPI + metformin group

SUMMARY:
This is a single-center, randomized controlled clinical trial with a parallel-group design conducted at Minia University hospital.

DETAILED DESCRIPTION:
All patients admitted to Diabetes clinics of Minia University Hospital, will be screened for the eligibility criteria.

diabetic patients (aged above 50 years) with uncontrolled diabetes on oral hypoglycemic drugs. 105 patients will be enrolled and randomized into three groups.

Group I=35 T2DM patients given DPP4Is Group II=35 T2DM patients given DPP4Is and metformin. Group III=35 patients will be given placebo (only adjust their drugs to control blood glucose level)

ELIGIBILITY:
Inclusion Criteria:

Type-2 diabetic adult subjects (above 50 years old) who had uncontrolled (A1c=8-9 %) blood glucose levels with an oral hypoglycemic drug at the screening visit were eligible to participate.

Exclusion Criteria:

Those with type1 diabetes or ketoacidosis, end organ failure as chronic renal failure (estimated serum creatinine level ≥ 1.5mg/dl in male and ≥ 1.4mg/dl in female), liver cell failure (elevated alanine transaminase (ALT) and aspartate transaminase (AST) ≥ 2 folds), and heart failure, previous history of pancreatitis, and pregnant or lactating females were excluded from the study.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Serum Inflammatory mediators; TNF-α | Before and post 6 month of treatment
  ELISA kits
MMSE score | Before and post 6 month of treatment
  Validated questionnaire assessing the Estimation of Mini Mental State The MMSE has a maximum score of 30 points. The scores are generally grouped as follows: 25-30 points: normal cognition 21-24 points: mild dementia 10-20 points: moderate dementia Examination (MMSE) score
PHQ-9 | Before and post 6 month of treatment
  Validated questionnaire assessing patient mental health and depression PHQ-9 scores of 5, 10, 15, and 20 represents mild, moderate, moderately severe and severe depression.;
serum amyloid-β | Before and post 6 month of treatment

SECONDARY OUTCOMES:
Serum Insulin | Before and post 6 month of treatment
  ElISA kits
Serum fasting and 2-he post prandial glucose | Before and post 6 month of treatment
HOMA-IR | Before and post 6 month of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University hospital, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided